CLINICAL TRIAL: NCT03162146
Title: Influence of Medical and Nursing Teams Composition on Patient Mortality in Intensive Care
Brief Title: Team Elements Associated With Mortality in Intensive Care
Acronym: TEAMIC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0031
Record Dates: First submitted 2017-05-17; First posted 2017-05-22 (Actual); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Intensive Care Unit Stay; Death
MeSH Terms: conditions — Death | interventions — Death Domain; Intensive Care Units

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient admitted to intensive care unit: All patients requiring intensive care unit stay
  Interventions: Other: Deaths in intensive care unit

INTERVENTIONS:
Other: Deaths in intensive care unit — Assessment of the influence of team familiarity among the members of medical and nursing staffs on risk of patient death

SUMMARY:
The individual characteristics and interactions of health care workers in intensive care units may influence patient safety. This study aims to quantify the influence of team familiarity among the members of medical and nursing staffs on risk of patient death.

ELIGIBILITY:
Inclusion Criteria:

* All patients who were admitted to 9 French intensive care units from January 1st 2011 to December 31st 2016

Exclusion Criteria:

* Patients admitted in pediatrics intensive care units and in specialized burns units

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient admitted to intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 43378 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Patient mortality | At the time of intensive care unit discharge up to a maximum of 6 years since admission
  Mortality with stratification on patients for whom a forego life-sustaining therapy decision was made

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Réanimation médicale, Hôpital de la Croix Rousse, Lyon, France

IPD SHARING:
Plan to Share IPD: No